CLINICAL TRIAL: NCT01119794
Title: Ofatumumab in Combination With Bortesomib in Patients With Relapsed or Refractory Low-Grade Non-Hodgkins Lymphoma
Brief Title: Ofatumumab and Bortezomib for Patients With Low-grade B-cell Non-hodgkin Lymphoma That Relapse After Rituximab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other); Memorial Hospital of Rhode Island (Other); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Eric Winer, MD, PI, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG-NHL-227
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Results first posted 2015-08-11 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Lymphoma, Non-Hodgkins
Keywords: B-cell small lymphocytic lymphoma; marginal zone lymphoma; follicular lymphoma; mantle cell lymphoma; Waldenström macroglobulinemia.; Low Grade B cell Non-Hodgkins Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia | interventions — ofatumumab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ofatumumab and bortezomib (Experimental): Ofatumumab 1000 mg IV Cycle 1 on day 1, 8, 15 and 22 Bortezomib 1.6 mg/m2 IV Ofatumumab 1000 mg IV on day 1 maintenance phase Patients will remain until progression
  Interventions: Drug: Ofatumumab and Bortezomib

INTERVENTIONS:
Drug: Ofatumumab and Bortezomib — Ofatumumab 1000 mg IV Cycle 1 on day 1, 8, 15 and 22 Bortezomib 1.6 mg/m2 IV Ofatumumab 1000 mg IV on day 1 maintenance phase Patients will remain until progression

SUMMARY:
The purpose of this study is to: Investigate the Overall Response Rate (ORR) of the combination of ofatumumab and bortezomib in patients with low-grade B-cell non-Hodgkin lymphoma (LG-NHL) that relapse beyond 6 months of a previous rituximab-containing regimen.

DETAILED DESCRIPTION:
41 patients will be enrolled in this trial with low grade lymphomas and will be given Ofatumumab 1000 mg and Bortezomib IV 1.6 mg/m2 weekly times 4 treatments and will then receive maintenance treatment with the 2 agents every 2 months for 1 year unless disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients are required to have histologically confirmed lymphoma according to the WHO/Revised European-American Lymphoma classification, including B-cell small lymphocytic lymphoma (SLL); marginal zone lymphoma (MZL); follicular lymphoma (FL), grades 1, 2, or 3; mantle cell lymphoma (MCL); and Waldenström macroglobulinemia. Prior history of transformed lymphoma is permitted as long as recent biopsies revealed no evidence of aggressive lymphoma and it has been > 3years since prior aggressive lymphoma
* Patients must measurable disease (defined as 1 cm with spiral computed tomography scan)
* Relapse of disease beyond 6 months after rituximab-containing regimen
* Patients had to have received no more than three prior lines of conventional cytotoxic therapy, and were required to have stopped receiving cytotoxic chemotherapy for at least 4 weeks before study enrollment
* Absolute neutrophil count > 1,500/uL and Platelet > 100,000/uL (if known lymphomatous involvement of the bone marrow, then absolute neutrophil count > 750/uL and platelet count of > 50,000/uL) within 14 days of enrollment.
* Total bilirubin < 1.5 x upper institutional limit of normal (ULN), and AST or ALT < 2.5 x ULN (< 3 x ULN if the patient had liver involvement); alkaline phosphatase < 2.5x upper limit of normal; and a creatinine < 2mg/dl within 14 days of enrollment.
* ECOG performance status 0 to 2
* Minimum life expectancy of 6 months
* Age older than 18 years
* Voluntary, signed written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.

Exclusion Criteria:

* Subjects who have current active hepatic or biliary disease asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Documented infection with HIV
* Positive serology for Hepatitis B defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HB DNA test will be performed and if positive the subject will be excluded.
* Central nervous system or meningeal involvement by lymphoma
* Prior transplantation
* Contraindication to any drug contained in the chemotherapy regimens
* Any serious active disease or co-morbid condition that would impair protocol treatment.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal call carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Prior treatment with any anti-CD20 monoclonal antibody, with the exception of rituximab, or any proteasome inhibitor.
* Patient has Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to boron or mannitol.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum pregnancy test result obtained during screening. A pregnancy test must be performed within 7 days prior to study drug. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs within 4 weeks before enrollment or 5 half lives of the investigational agent.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Castillo, MD, Principal Investigator — Lifespan
Locations (3):
- United States (3):
  - Dartmouth-Hitchcock Medical Center, Hanover, New Hampshire
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- Ofatumumab IV,: Ofatumumab 1000 mg IV Cycle 1 on day 1, 8, 15 and 22,
  Ofatumumab and Bortezomib: Ofatumumab 1000 mg IV Cycle 1 on day 1, 8, 15 and 22- in the induction phase Ofatumumab 1000 mg IV on day 1- will receive in the maintenance phase Patients will remain until progression
Period: Overall Study
Arm/Group | Ofatumumab IV,
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab IV,
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 68 [55 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) of the Combination of Ofatumumab and Bortezomib in Patients Receiving Study Treatment
Description: Response was assessed based on Bone marrow biopsy and CT scan. Best responses are used for Response Rate and CR and PR only.
  Complete Response - CR:
  • Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy.
  Partial Response - PR:
  • At least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses.
  Stable Disease - SD:
  • A patient is considered to have SD when he or she fails to attain the criteria needed for a CR or PR, but does not fulfill those for progressive disease
  Relapsed Disease:
  • Lymph nodes should be considered abnormal if the long axis is more than 1.5 cm regardless of the short axis.
Time Frame: Bone Marrow Biopsy: Every 2 months for 1 year then every 4 months until progression for approximately 1 year/Via CT scan: every 4 months until progression, for a total of approximately 2 years
Population: 8/10 patients were evaluable as 2 withdrew
Measure: Number; unit: participants
Arm/Group | Ofatumumab IV,
Number analyzed (Participants) | 8
participants
  CR | 2
  PR | 1
  SD | 3
  Progression | 2

ADVERSE EVENTS:
Arm/Group | Ofatumumab IV,
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ofatumumab IV, (N=10)
diarrhea (Gastrointestinal disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1)
nausea (Investigations) | 1 (1)
vomitting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ofatumumab IV, (N=10)
infusion reaction (Investigations) | 7 (7)
diarrhea (Gastrointestinal disorders) | 4 (4)
glucose (Investigations) | 6 (6)
abdominal pain (Investigations) | 1 (1)
nausea (Investigations) | 3 (3)
shortness of breath (Investigations) | 2 (2)
edema (Investigations) | 3 (3)
fatigue (Investigations) | 4 (4)
white blood cell decrease (Investigations) | 2 (2)
general pain (General disorders) | 2 (2)
rash (Investigations) | 3 (3)
derm skin other (Investigations) | 2 (2)
anemia (Investigations) | 6 (6)
thrombocytopenia (Investigations) | 5 (5)
neuropathy (Investigations) | 2 (2)
constipation (Gastrointestinal disorders) | 1 (1)
neutropenia (Investigations) | 1 (1)
Red blodd cell (Investigations) | 2 (2)
Lymphopenia (Investigations) | 4 (4)
hyponatremia (Investigations) | 2 (2)
Liver function test abnormalities (Investigations) | 2 (2)
muscle aches (General disorders) | 1 (1)
phosphorus (Investigations) | 2 (2)
sweating (Investigations) | 1 (1)
mood alteration (Psychiatric disorders) | 1 (1)
phlebitis (Investigations) | 1 (1)
creatinine (Investigations) | 1 (1)
dehydration (Investigations) | 1 (1)
hip pain (Investigations) | 1 (1)
cough (Investigations) | 1 (1)
back pain (Investigations) | 1 (1)
heartburn (Investigations) | 1 (1)
upper respiratory infection (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No